CLINICAL TRIAL: NCT06285188
Title: Immunomonitoring of Mold Invasive Infections
Acronym: IMMUNOFIL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221174; 2023-A01398-37 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Invasive Fungal Disease; Mold Invasive Fungal Infection: Aspergillus, Mucorales, Fusarium, Scedosporium
Keywords: Invasive fungal diseases,; adaptative immunity against filamentous fungi; immune checkpoint molecules; anti-PD1
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of patients with mold invasive fungal infection: Patients >18 y, with a diagnosis of proven or probable mold invasive fungal infection (Aspergillus, Mucorales, Fusarium or Scedosporium), according to modified 2019 EORTC/MGS criteria, at diagnosis or at a refractory state after a first-line antifungal treatment

SUMMARY:
Mold invasive infections are associated with an important mortality despite optimization of the antifungal treatment. In a few case reports, immune checkpoints inhibitors, initially developed for neoplastic diseases, have shown a potential beneficial effect in such devastating infections by restoring an efficient immune response. The investigators propose a longitudinal monitoring of the adaptative immune response, notably immune checkpoint expression on T cells, during mold invasive infections to help identify the patients who could benefit from the adjunction of immunotherapy and the optimal timing of such strategy.

DETAILED DESCRIPTION:
Invasive fungal diseases (IFD) still cause substantial morbidity and mortality. New therapeutic approaches are therefore urgently needed, notably for patients not responding to conventional antifungal treatment. One strategy to prevent treatment failure is to improve the immune functions of immunocompromised hosts. Indeed, antifungals therapeutic efficacy is limited without the help of host immune reactivity (Stevens et al., 2000). As several studies have suggested that IFD are associated with an impaired Th1 host immune response, various cytokines have been evaluated in experimental and human fungal infections. In particular, adjunction of recombinant IFNγ has been proposed as a treatment option in patients with poor prognosis IFD with partial success. More recently, it has been shown that, when T cells are exposed to persistent antigens and/or inflammatory signals due to inefficient control of persisting infections, or in the context of tumors, a deterioration of their functions is observed, a state called "exhaustion". Molecular pathways involved in exhaustion have been partially deciphered, highlighting the importance of molecules called immune checkpoint such as PD-1 or CTLA-4. Furthermore, it was shown that blockade of these molecules can reverse this dysfunctional state. Immune checkpoint inhibitors (such as anti-PD1 antibodies) have become major weapons in oncology. In infectious diseases, and more particularly IFDs, data are much more limited. In animal models of several IFD, such as aspergillosis, cryptococcosis and histoplasmosis, repetitive administration of anti-PD-1 monoclonal antibodies significantly improved fungal clearance and survival of lethally infected animals. In humans, three case-reports, including one published by our team, have reported the efficacy of anti-PD-1 therapy combined with IFN-γ in the treatment of refractory IFDs. Therefore, by reversing T cell exhaustion, immune checkpoint blockade represents a therapeutic perspective for IFD treatment.

The use of immune checkpoint inhibitors may, however, entail severe, notably autoimmune off-target adverse effects and should be carefully balanced and monitored. The development of tools allowing identification of patients who could benefit from immunotherapy is of particular importance as well as assessment of the optimal timing of these innovative treatments. As such, a better understanding of the host immune response is one of the major approaches to developing new or improved antifungal strategies to control IFDs. Longitudinal data regarding the evolution of exhaustion markers expression in T cells of patients treated for an IFD are lacking.

The goal is to better characterize the adaptative immune response directed against molds, notably immune checkpoint expression, in order to identify the patients who could benefit from the adjunction of immunotherapy and the optimal timing of such strategy.

For this purpose, the investigators will include adult patients with mold IFD either at diagnosis or refractory to conventional therapy. They will measure activation and exhaustion markers on circulating T cells and monocytes by flow cytometry at three timepoints (enrollment, day 14 and week 6). Moreover, for patients with invasive aspergillosis or mucormycosis, they will evaluate the capacity of specific T cells to produce Th1, Th2 and Th 17 cytokines and to proliferate after specific antigenic stimulation, in the absence and in the presence of an anti-PD1 antibody in vitro (4 colors FLUOROSPOT) at two timepoint (enrollment and week 6). These data will provide a longitudinal assessment of the anti-fungal immune response. They will be correlated with the underlying diseases of the patients, the type of mold infection (aspergillosis, mucormycosis, fusariosis or scedosporiosis), the treatment received and the outcome. These results should help to better identify patients who could benefit from adjunctive anti PD-1 treatment and the optimal timing for such treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mold invasive fungal infection: Aspergillus, Mucorales, Fusarium, Scedosporium
* Proven or probable according to 2019 EORTC/MGS criteria modified by the adjunction of diabetes mellitus in the host criteria and Mucorales PCR in the microbiological criteria
* Within 14 days of IFD diagnosis or
* a refractory state defined by the 2009 MGS/EORT failure criteria (clinical, radiological, or microbiological failure) of a first-line antifungal treatment leading to a change of therapy by the attending physician of the patient
* Patients with aspergillosis or mucormycosis for whom ELISPOTs are developed: Total lymphocyte count > 700/mm3 on the last sample taken
* No opposition to participate to the research
* Affiliated or beneficiary of social security system

Exclusion Criteria:

* Bacterial co-infection in the last 14 days
* Previous treatment with anti-PD1 antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care centers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Immune checkpoint expression on T cells | Day 0, day 14, week 6
  percentage of circulating T cells expressing immune checkpoint molecules as well as the intracellular transcription factor TCF1 and mean fluorescence intensity (MFI) of this expression in each cell sub-population

SECONDARY OUTCOMES:
Aspergillus/Mucorales FLUOROSPOT | Day 0, week 6
  Qualitative and quantitative measure of specific T cells IFN-γ/IL-2/IL-5/IL-17 production by FLUOROSPOT after antigenic stimulation in absence and presence of an anti-PD1 antibody in patients with invasive aspergillosis or mucormycosis
T cell proliferation | Day 0, week 6
  T cell proliferation test after antigenic stimulation
Immune checkpoint expression on monocytes | Day 0, day 14, week 6
  Percentage of circulating monocytes expressing immune checkpoint molecules

CONTACTS AND LOCATIONS:
Overall Officials: Fanny LANTERNIER, MD, PhD, Study Chair — APHP
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No